CLINICAL TRIAL: NCT06557837
Title: Evaluation of Deterioration in Body Posture of Older Patients During Gait Compared to Stance
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: AO Foundation, AO Spine (Other)
Responsible Party: Principal Investigator, Armand Dominik Škapin, Principal Investigator, University Medical Centre Ljubljana
Other Study IDs: 0120-22/2023/47; AOS-Startup-23-028 (Other Grant/Funding Number: AO Spine)
Record Dates: First submitted 2024-08-07; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Degenerative Spine Disease; Sagittal Balance
MeSH Terms: interventions — Pain Measurement; Muscle Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with sagittal imbalance: Patients that have pelvic incidence-lumbar lordosis deficit (PI-LL) greater than 10 or sagittal vertical axis (SVA) greater than 4 centimetres on X-ray imaging.
  Interventions: Diagnostic Test: Questionnaires and pain assessment; Diagnostic Test: Standing sagittal whole spine X-ray; Diagnostic Test: Dynamic test; Diagnostic Test: Muscle strength and body composition measurement
- Control group: Participants with normal pelvic incidence-lumbar lordosis deficit (PI-LL) and sagittal vertical axis (SVA) on X-ray imaging.
  Interventions: Diagnostic Test: Questionnaires and pain assessment; Diagnostic Test: Standing sagittal whole spine X-ray; Diagnostic Test: Dynamic test; Diagnostic Test: Muscle strength and body composition measurement

INTERVENTIONS:
Diagnostic Test: Questionnaires and pain assessment — Participants complete two questionnaires: the Oswestry Disability Index (ODI) and the EQ-5D-5L. They also rate their low back pain using the Visual Analogue Score (VAS) scale and respond to two additional questions about their posture and gait.
Diagnostic Test: Standing sagittal whole spine X-ray — Participants undergo standard preoperative X-ray imaging of the entire spine to capture the upright posture. This imaging is conducted before and after 6-minute of continuous walking to compare changes in spino-pelvic and sagittal balance parameters.
Diagnostic Test: Dynamic test — With the dynamic test, we analyze body movements of participants during gait using 49 reflective markers placed on their bodies according to the Qualisys PAF package: Instituti Ortopedici Rizzoli (IOR) and 10 EMG electrodes on specific leg and back muscles. Participants walk for 6 minutes between two cones set 7 meters apart, while a 12-camera Qualisys Motion Capture System tracks marker movements for comprehensive kinematic analysis. Data are recorded at five key moments: standing before and after the test, and during three phases of gait (at the beginning, middle, and end). Participants are barefoot and dressed in underwear for accurate measurement. Static recordings before and after walking involve stepping on a tensiometric force plate to measure the center of gravity. Before the test, participants perform stretching exercises to ensure consistent preparation.
Diagnostic Test: Muscle strength and body composition measurement — Participants have their body composition analyzed and the maximum isometric strength of their paraspinal and abdominal muscles measured using the Dr. Wolff BackCheck device.

SUMMARY:
The goal of this observational study is to analyze how spinal alignment changes when walking compared to standing still in adults aged 50 to 80 years who have sagittal imbalance. The main questions we aim to answer are:

1. Do patients with radiological parameters indicative of sagittal imbalance experience a statistically significant deterioration in sagittal balance during walking compared to a control group?
2. Do radiographs taken after six minutes of walking provide comparable results to dynamic measurements during the walking test?
3. Do patients with a greater deterioration in sagittal balance during walking show poorer clinical self-assessment scores?
4. Is there a significant correlation between parameters obtained using established diagnostic methods and the degree of sagittal balance deterioration during walking?

Participants will be divided into two groups: patients with radiological indicators of sagittal imbalance and a control group of healthy individuals with back pain of similar age. Participants will:

1. Complete questionnaires about their back pain and mobility.
2. Have X-ray images taken of their spine before and after walking for six minutes.
3. Undergo muscle strength tests and gait analysis using motion capture and electromyography (EMG) to monitor muscle activity while walking.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic incidence-lumbar lordosis deficit (PI-LL) greater than 10 or sagittal vertical axis (SVA) greater than 4 centimeters
* The main symptom is low back pain
* Age between 50-80 years.

Exclusion Criteria:

* Symptoms of spinal stenosis
* Previous instrumented spinal surgery
* Cobb angle greater than 30°
* Symptoms of hip or knee arthrosis
* Symptoms of vascular intermittent claudication
* Cardio-pulmonary disease that lowers the patient's physical capability
* Neuromuscular disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are selected from the outpatient clinic at the specialized orthopedic department of the University Medical Centre Ljubljana.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in C7-STS During Gait | Within 2 months from enrollment
  The change in the value of the C7 - sagittal trunk shift (C7-STS) will be measured at five points during the dynamic test. The measurement is in millimeters. C7-STS is defined as the distance between vertical line through the marker placed on spinous process C7 and the marker on spinous process L5.
Change in AM-STS During Gait | Within 2 months from enrollment
  The change in the value of the Auditory meatus - sagittal trunk shift (AM-STS) will be measured at five points during the dynamic test. The measurement is in millimeters. AM-STS is defined as the distance between vertical line through the middle of the markers placed on each side of the head just above the ear and the middle of the markers placed on both greater trochanters.
Change in SVA on X-ray During Walking | At enrollment
  A comparison of the Sagittal Vertical Axis (SVA) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in millimeters. SVA is measured as the horizontal distance between a vertical line from the center of the C7 vertebra and the posterior superior corner of the sacrum on a sagittal X-ray.
Change in CAM-HA on X-ray During Walking | At enrollment
  A comparison of the Center of Auditory Meatus to Hip Axis Plumbline (CAM-HA) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in millimeters. CAM-HA is measured as the horizontal distance between a vertical line from the center of auditory meatus and the axis of the femoral heads on a sagittal X-ray.

SECONDARY OUTCOMES:
Change in PA During Gait | Within 2 months from enrollment
  The change in the value of the Pelvic angle (PA) will be measured at five points during the dynamic test. The measurement is in degrees. PA is defined as the angle between the markers placed on the posterior superior iliac spines and anterior superior iliac spines and horizontal plane.
Change in LLA During Gait | Within 2 months from enrollment
  The change in the value of the Lumbar lordosis angle (LLA) will be measured at five points during the dynamic test. The measurement is in degrees. LLA is defined as the angle between the markers placed on spinous processes of L1, L3 and L5.
Change in TKA During Gait | Within 2 months from enrollment
  The change in the value of the Thoracic kyphosis angle (TKA) will be measured at five points during the dynamic test. The measurement is in degrees. TKA is defined as the angle between the markers placed on spinous process of C7, spinous process of vertebra between the inferior edge of the scapulae and spinous process L1.
Change in STA During Gait | Within 2 months from enrollment
  The change in the value of the Sagittal trunk angle (STA) will be measured at five points during the dynamic test. The measurement is in degrees. STA is defined as the angle between the line connecting the middle of the markers placed on each side of the head just above the ear and the middle of the markers placed on both greater trochanters and vertical line.
Change in GTA During Gait | Within 2 months from enrollment
  The change in the value of the Global tilt angle (GTA) will be measured at five points during the dynamic test. The measurement is in degrees. GTA is defined as the angle between the markers placed on spinous process C7, L5 and the middle of the markers placed on both greater trochanters.
Change in PT on X-ray During Walking | At enrollment
  A comparison of the Pelvic Tilt (PT) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in degrees. PT is defined as the angle between the vertical and the line connecting the center of the sacral endplate to the axis of the femoral heads on a sagittal X-ray.
Change in SS on X-ray During Walking | At enrollment
  A comparison of the Sacral Slope (SS) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in degrees. SS is defined as the angle between a line tangent to the upper S1 endplate and horizontal line.
Change in LL on X-ray During Walking | At enrollment
  A comparison of the Lumbar Lordosis (LL) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in degrees. LL is defined as the angle between the superior endplate of the first lumbar vertebra and the superior endplate of the first sacral vertebra.
Change in TK on X-ray During Walking | At enrollment
  A comparison of the Thoracic Kyphosis (TK) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in degrees. TK is defined as the angle between the superior endplate of the first thoracic vertebra and the inferior endplate of the twelfth thoracic vertebra.
Change in PI-LL on X-ray During Walking | At enrollment
  A comparison of the Pelvic Incidence-Lumbar Lordosis Deficit (PI-LL) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in degrees. PI-LL is defined as the difference between the pelvic incidence (PI) and lumbar lordosis (LL) angles.
Change in Angle of the hip on X-ray During Walking | At enrollment
  A comparison of the Angle of the Hip in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in degrees. Angle of the Hip is defined as the angle between the line connecting the center of the sacral endplate to the axis of the femoral heads and the line drawn from the axis of the femoral heads along the femoral shaft.
Change in OD-HA on X-ray During Walking | At enrollment
  A comparison of the Odontoid Hip Axis Angle (OD-HA) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in degrees. OD-HA is defined as the angle between the vertical and the highest point of the odontoid process (dens) connecting to the center of the acetabulum (bi-coxo-femoral axis).
Change in GT on X-ray During Walking | At enrollment
  A comparison of the Global Tilt (GT) in an upright stance, as captured by X-ray imaging, before and after 6 minutes of continuous walking. The measurement is in degrees. GT is defined as the angle between a vertical line and a line drawn from the center of the C7 vertebra to the center of the sacral endplate.
Oswestry Disability Index (ODI) Questionnaire | At enrollment
  The Oswestry Disability Index (ODI) is a questionnaire used to assess a patient's level of disability related to lower back pain. It is scored on a scale from 0 to 100%, where higher scores indicate worse outcomes.
EQ-5D-5L Questionnaire | At enrollment
  The European Quality of Life in 5 Dimensions and 5 Levels (EQ-5D-5L) is a standardized questionnaire used to measure a patient's health-related quality of life across five dimensions and five levels. It is scored on a scale from -0,573 to 1, where higher scores indicate better outcomes.
Visual Analogue Score (VAS) for low back pain | At enrollment
  The Visual Analogue Score (VAS) for low back pain is a tool used to measure patient's pain intensity in the lower back. It is scored on a scale from 0 to 10, where higher scores indicate worse outcomes.
Additional Question: Is it hard for you to stand upright? | At enrollment
  The additional question "Is it hard for you to stand upright?" is assessed with a "yes" or "no" response, where "yes" indicates a worse outcome, signifying difficulty in maintaining an upright posture.
Additional Question: Does your body lean forward during gait? | At enrollment
  The additional question "Does your body lean forward during gait?" is assessed with a "yes" or "no" response, where "yes" indicates a worse outcome, signifying a forward lean during walking.
Maximum Isometric Strength of the Paraspinal Muscles | Within 2 months from enrollment
  The maximum isometric strength of the paraspinal muscles is measured using the Dr. Wolff BackCheck device. The muscle strength is recorded in Newton-meters (Nm) and then adjusted according to the participant's body weight for accurate comparison.
Maximum Isometric Strength of the Abdominal Muscles | Within 2 months from enrollment
  The maximum isometric strength of the abdominal muscles is measured using the Dr. Wolff BackCheck device. The muscle strength is recorded in Newton-meters (Nm) and then adjusted according to the participant's body weight for accurate comparison.
Skeletal Muscle Mass | Within 2 months from enrollment
  Patients have their skeletal muscle mass measured using the InBody 720 device, with the results recorded in kilograms (kg).
Body Fat Mass | Within 2 months from enrollment
  Patients have their body fat mass measured using the InBody 720 device, with the results recorded in kilograms (kg).
Body Fat Percentage | Within 2 months from enrollment
  Patients have their body fat percentage measured using the InBody 720 device, with the results recorded as a percentage (%).
Total Body Water | Within 2 months from enrollment
  Patients have their total body water measured using the InBody 720 device, with the results recorded in liters (L).
Extracellular Water / Total Body Water | Within 2 months from enrollment
  Patients have their extracellular water versus total body water proportion measured using the InBody 720 device, with the results recorded as a ratio.

CONTACTS AND LOCATIONS:
Locations (2):
- Slovenia (2):
  - Faculty of Sport, University of Ljubljana, Ljubljana
  - University Medical Centre Ljubljana, Ljubljana

IPD SHARING:
Plan to Share IPD: No